CLINICAL TRIAL: NCT04007991
Title: Multicenter, Placebo-Controlled, Double-Blind, Randomized, Parallel-Group, Phase 2b Study to Evaluate the Efficacy and Safety of Ecopipam in Children and Adolescents With Tourette's Syndrome
Brief Title: Ecopipam Tablets to Study Tourette's Syndrome in Children and Adolescents
Acronym: D1AMOND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emalex Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EBS-101-CL-001
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — ecopipam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ecopipam HCI 2 mg/kg/day (Experimental): Ecopipam HCl 12.5-, 50-, 75- and 100-mg tablets; 2 mg/kg/day target dose; oral administration daily in evenings
  Interventions: Drug: Ecopipam
- Placebo (Placebo Comparator): Matching Placebo tablets taken orally in the evening
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ecopipam — Ecopipam HCI tablets administered PO to establish 2 mg/kg/day
  Arms: Ecopipam HCI 2 mg/kg/day
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
This study evaluates the effect of ecopipam tablets in children and adolescents in the treatment of Tourette's Syndrome (TS). Half of the participants will receive ecopipam tablets, while the other half will receive matching placebo tablets

DETAILED DESCRIPTION:
Multicenter, placebo-controlled, double-blind, randomized, parallel-group, Phase 2b study in pediatric subjects (aged greater than equal to 6 to less than 18 years of age) with TS. Following a 28-day Screening period and Baseline visit, eligible subjects will be randomized 1:1 to receive either ecopipam hydrochloride (HCl) or matching placebo for a 12 week treatment period. Doses will be titrated up and down from target dose of 2 mg/kg/day. Follow Up visit will be conducted after the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 6 and < 18 years of age
* ≥ 18 kg (~ 40 lbs.)
* TS diagnosis and both motor and vocal tics that cause impairment with normal routines
* Minimum score of 20 on the YGTSS-Total Tic Score
* May not be taking any medications used to treat motor or vocal tics for at least 14 days prior to Baseline.
* Effective contraception during the study and 30 days after last study dose for sexually active subjects

Exclusion Criteria:

* Certain mood or psychiatric disorders (i.e., dementia, bipolar disorder, schizophrenia, major depressive disorder)
* Unstable medical illness or clinically significant lab abnormalities
* Risk of suicide
* Pregnant or lactating women
* Moderate to severe renal insufficiency
* Hepatic insufficiency
* Positive urine drug screen
* Unstable doses for drugs to treat anxiety, depression, Attention Deficit Hyperactivity Disorder
* Certain medications that would lead to drug interactions
* Recent behavioral therapy

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 153 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (70):
- United States (53):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Advanced Research Center Inc., Anaheim, California
  - UCLA, Los Angeles, California
  - PCSD-Feighner Research, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Yale School of Medicine, New Haven, Connecticut
  - Sarkis Clinical Trials, Gainesville, Florida
  - Northwest Florida Clinical Research Group, LLC, Gulf Breeze, Florida
  - Research in Miami Inc., Hialeah, Florida
  - University of Miami, Miami, Florida
  - MedBio Trials, North Miami, Florida
  - APG Research LLC, Orlando, Florida
  - University of South Florida, St. Petersburg, Florida
  - Pediatric Epilepsy and Neurology Specialists, Tampa, Florida
  - Pediatric Neurology, PA, Winter Park, Florida
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - The University of Chicago Hospitals, Chicago, Illinois
  - AMR - Baber Research Inc., Naperville, Illinois
  - Psychiatric Associates, Overland Park, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Michigan Clinical Research Institute PC, Ann Arbor, Michigan
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - Helen DeVos Children's Hospital / Spectrum Health Medical Group, Wyoming, Michigan
  - St. Charles Psychiatric Associates dba Midwest Research Group, Saint Charles, Missouri
  - Movement Disorders Center, St Louis, Missouri
  - Alivation Research, LLC, Lincoln, Nebraska
  - Center for Psychiatry and Behavioral Medicine Inc., Las Vegas, Nevada
  - The NeuroCognitive Institute, Mount Arlington, New Jersey
  - Clinical Research Center of NJ, Voorhees Township, New Jersey
  - New York Neurology Associates P.C, New York, New York
  - Hapworth Research Inc., New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Mood Disorders Consulting Medicine PLLC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Quest Therapeutics of Avon Lake, Avon Lake, Ohio
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - North Star Medical Research LLC, Middleburg Heights, Ohio
  - Suburban Research Associates, Media, Pennsylvania
  - Coastal Pediatric Research, Charleston, South Carolina
  - Access Clinical Trials, Inc., Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Clinical Trials LLC, Bellaire, Texas
  - Relaro Medical Trials, Dallas, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Road Runner Research Ltd., San Antonio, Texas
  - Noetic Psychiatry, Springville, Utah
  - University of Virginia, Charlottesville, Virginia
  - Eastside Therapeutic Resource Inc dba Core Clinical Research, Everett, Washington
- Canada (3):
  - The Kids Clinic Inc, Ajax, Ontario
  - Center for Pediatric Excellence, Ottawa, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
- France (2):
  - CHU Poitiers, Poitiers
  - Hopital Robert Debre, Paris, Île-de-France Region
- Germany (5):
  - Psychiatric Clinic of Ludwig Maximilians Universitaet Muenchen, Munich, Bavaria
  - Department of Psychiatry, Socialpsychiatry and Psychotherapy, Hannover Medical School, Hanover, Lower Saxony
  - Dept. Child Adolescent Psychiatry Uni. Freiburg, Freiburg im Breisgau
  - Zentralinstitut fuer Seelische Gesundheit, Mannheim
  - Pharmakologisches Studienzentrum Chemnitz GmbH, Mittweida
- Poland (7):
  - Gdanskie Centrum Zdrowia Sp z o.o., Gdansk
  - Centrum Bada Klinicznych PI-House Sp. z o.o., Gdansk
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - NZOZ Wielospecjalistyczna Poradnia Lekarska Synapsis, Katowice
  - Centrum Medyczne Plejady, Krakow
  - Wojewdzki Specjalistyczny Szpital Dziecicy im. sw. Ludwika w Krakowie, Krakow
  - Med-Polonia Sp. z o. o., Poznan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 45 sites in 5 countries (United States, Canada, Germany, France, and Poland) from 28 June 2019 (first participant first visit) and 23 September 2021 (last participant last visit).
Pre-assignment Details: A total of 215 participants were screened, of which 61 participants were screen failures and 153 participants were randomized in 1:1 ratio to receive ecopipam HCl and placebo.
Groups:
- Ecopipam HCI 2 mg/kg/Day: Participants received a targeted steady-state dose of 2 milligram per kilogram per day (mg/kg/day) of ecopipam HCl tablets orally, once daily during a titration and treatment period for a total of 12 weeks.
- Placebo: Participants received matching placebo tablets orally, once daily during a titration and treatment period for a total of 12 weeks.
Period: Overall Study
Arm/Group | Ecopipam HCI 2 mg/kg/Day | Placebo
Started | 76 | 77
Safety Set (The Safety Set (SS) included all participants who received at least one dose of study drug.) | 76 | 77
The Modified Intention-to-Treat Set (The Modified Intention-to-Treat (mITT) set included all randomized participants who received at least one dose of study drug and had at least 1 post-baseline scoring of the YGTSS (Yale Global Tic Severity Scale).) | 74 | 75
Completed | 66 | 71
Not Completed | 10 | 6
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Non-compliance with Study Drug | 0 | 1
Not completed — Withdrawal by Parent/Caregiver | 1 | 2
Not completed — Adverse event, non-fatal | 5 | 0
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Set included all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ecopipam HCI 2 mg/kg/Day | Placebo | Total
Number analyzed (Participants) | 76 | 77 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.6 (2.78) | 12.6 (2.63) | 12.6 (2.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 24 | 41
  Male | 59 | 53 | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 11 | 24
  Not Hispanic or Latino | 63 | 66 | 129
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 66 | 72 | 138
  Black or African American | 6 | 3 | 9
  Asian | 1 | 2 | 3
  American Indian or Alaska Native | 1 | 0 | 1
  Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Yale Global Tic Severity Scale-Total Tic Score (YGTSS-TTS) at Week 12
Description: The YGTSS was a semi-structured clinical interview designed to measure the tic severity. This scale consisted of a tic inventory, with 5 separate rating scales to rate the severity of symptoms, and an impairment ranking. Ratings were made along 5 different dimensions on a scale of 0=none to 5=severe for motor and vocal tics, each including number, frequency, intensity, complexity, and interference. The YGTSS TTS was the summation of the severity scores of motor and vocal tics. The total tic score (TTS) ranged from 0 (none) to 50 (severe) with higher score represent more severe symptoms. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12
Population: The mITT set included all randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline scoring of the YGTSS.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ecopipam HCI 2 mg/kg/Day | Placebo
Number analyzed (Participants) | 74 | 75
score on a scale | -9.87 (1.062) | -6.42 (1.006)
Statistical Analysis 1: Comparison: Ecopipam HCI 2 mg/kg/Day vs Placebo; Test type: Superiority; p = 0.011, ANCOVA — Change from baseline in YGTSS score as a continuous variable was based on mixed model for repeated measures (MMRM) analysis of covariance (ANCOVA) model with an unstructured covariance matrix; Difference in Least Square Mean = -3.44, 95% CI 2-sided [-6.09 to -0.79], Standard Error of Mean 1.351

2. Secondary Outcome: Change From Baseline in Clinical Global Impression of Tourette Syndrome Severity (CGI-TS-S) at Week 12
Description: Clinical Global Impression (CGI) scale was used to assess overall severity on a 7-point Likert scale consisted of 2 reliable and valid 7-item Likert scales used to assess severity and change in clinical symptoms. The CGI severity scale ranges from 1 = Normal, not at all ill; 2 = Borderline ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; 7 = Among the most extremely ill subject. 1 = "normal, not ill at all" to 7 = "extremely ill." A negative change indicates improvement in the condition.
Time Frame: Baseline, Week 12
Population: The mITT set included all randomized subjects who received at least 1 dose of study drug and had at least 1 post-baseline scoring of the YGTSS. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ecopipam HCI 2 mg/kg/Day | Placebo
Number analyzed (Participants) | 65 | 71
score on a scale | -0.91 (0.141) | -0.53 (0.130)

ADVERSE EVENTS:
Time Frame: Screening up to 30 days after the last dose ( up to Week 16)
Arm/Group | Ecopipam HCI 2 mg/kg/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/77
Serious Adverse Events (participants affected / at risk) | 2/76 | 1/77
Other Adverse Events (participants affected / at risk) | 47/76 | 38/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ecopipam HCI 2 mg/kg/Day (N=76) | Placebo (N=77)
Vomiting (Gastrointestinal disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Coronavirus infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ecopipam HCI 2 mg/kg/Day (N=76) | Placebo (N=77)
Contusion (Injury, poisoning and procedural complications) | 0 | 3
Fall (Injury, poisoning and procedural complications) | 2 | 0
Muscle strain (Injury, poisoning and procedural complications) | 2 | 0
Sunburn (Injury, poisoning and procedural complications) | 2 | 1
Headache (Nervous system disorders) | 12 | 7
Somnolence (Nervous system disorders) | 6 | 2
Dizziness (Nervous system disorders) | 3 | 0
Fatigue (General disorders) | 6 | 0
Pyrexia (General disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 4 | 0
Restlessness (Psychiatric disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 7 | 1
Depressed mood (Psychiatric disorders) | 3 | 2
Depression (Psychiatric disorders) | 1 | 2
Irritability (Psychiatric disorders) | 3 | 1
Middle insomnia (Psychiatric disorders) | 3 | 1
Sleep disorder (Psychiatric disorders) | 3 | 1
Tic (Psychiatric disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 5 | 4
Coronavirus infection (Infections and infestations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must consult their clinical trial agreement. In summary, PI shall have the right to publish, present or otherwise use the results for their research publication objectives, provided that such Publication does not disclose Confidential Information. PI shall submit in writing to Sponsor any material at least 90 days for review and comment. Sponsor shall advise PI of any information which is Confidential Information or which may impair Sponsor's ability to obtain patent protection.

DOCUMENTS (2):
  • Study Protocol (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT04007991/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/91/NCT04007991/SAP_001.pdf